CLINICAL TRIAL: NCT03348891
Title: TNF in Melanoma Patients Treated With Immunotherapy
Acronym: MELANFα
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17 CUTA 08
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Melanoma
Keywords: Melanoma; TNF; Immune checkpoints; Tumor-infiltrating lymphocytes; Cytokines; Circulating leukocytes
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subgroup 1 (Other): Patients treated with anti-PD-1 alone (nivolumab or pembrolizumab)
  Interventions: Other: Tumor biopsy specimens and blood samples
- Subgroup 2 (Other): Patients treated with the combined treatment anti-PD-1+anti-CTLA-4 (nivolumab + ipilimumab)
  Interventions: Other: Tumor biopsy specimens and blood samples

INTERVENTIONS:
Other: Tumor biopsy specimens and blood samples — Tumor biopsy specimens (if feasible) and blood samples will be collected at Baseline, Week 6 Day 1 (blood sample only) and Week 12 Day 1.

SUMMARY:
This trial is a translational proof-of-concept, open-label, prospective cohort study of 60 patients aiming to identify the clinical markers and/or biomarkers associated with therapeutic response to immune checkpoints inhibitors, in patients with advanced melanoma.

The study will be conducted on a population of patients treated with ICI in the context of routine care, separated in two subgroups:

* Subgroup 1: patients treated with anti-PD-1 alone (nivolumab or pembrolizumab)
* Subgroup 2: patients treated with the combined treatment anti-PD-1+anti-CTLA-4 (nivolumab + ipilimumab)

For each included patient, blood samples will be collected during baseline visit and during treatment period (at Week 6 Day 1 and Week 12 Day 1).

If feasible, tumor biopsy (of primary tumor or metastasis) will be performed during baseline and on Week 12 Day 1 visit (predose). If tumor biopsy is not feasible, available archived tumor specimen (frozen or FFPE block) may be collected for the study.

All included patients will be followed-up for tumor status and/or survival status every 3 months until a maximum duration of 1 year from the first study dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of study entry.
2. Patient with histologically-proven metastatic and/or unresectable melanoma (stage IIIc-IV, M1a-c as per AJCC 2009), including mucosal melanoma.
3. Patient for which a treatment with immune checkpoint inhibitor (nivolumab alone, pembrolizumab alone or nivolumab + ipilimumab) has been decided.
4. Subjects are included regardless of BRAFV600 mutation status. BRAFV600 mutation status must be documented.
5. Patient must be naïve to immune checkpoint inhibitor treatment for locally advanced and/or metastatic disease (i.e., no prior treatment with ICI and current treatment with ICI not yet started).
6. ECOG Performance status 0-2.
7. Life expectancy of at least 3 months.
8. Patient able to participate and willing to give informed consent prior to performance of any study-related procedures and to comply with the study protocol.
9. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Patient pregnant, or breast-feeding.
2. Uveal melanoma.
3. Any condition contraindicated with sampling procedures required by the protocol.
4. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.
5. Any current severe or uncontrolled disease, including, but not limited to ongoing or active infection.
6. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the discriminant capacity to predict progression at 12 weeks evaluated using RECIST V1.1 criteria. | 12 weeks per patient

SECONDARY OUTCOMES:
Objective response (i.e. complete or partial response) will be defined using RECIST V1.1 criteria at week 12. | 12 weeks per patient
Response duration is defined as the time from objective response until progression according to investigator judgment, or death. | 12 months per patient
Progression Free Survival is defined as the time from inclusion until progression according to investigator judgment, or death, whichever occurs first. | 12 months per patient
Immune related adverse event will be evaluated using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03. | 12 weeks per patient

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU Claude HURIEZ, Lille
  - CHU Montpellier Saint-Eloi, Montpellier
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse